CLINICAL TRIAL: NCT01921023
Title: An Open, Non-randomised, Study to Provide a Comparison of Data From a Conventional Blood Gas Analyser With Those Obtained From the CE Marked Proxima System
Brief Title: Comparison of Performance of a Conventional Blood Gas Analyser With the Proxima System
Status: Completed | Type: Observational
Sponsor: Sphere Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROX006
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-02

CONDITIONS: Analysis, Event History
Keywords: Blood Gas analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical investigation is being undertaken to examine the performance of the CE marked Proxima System - a patient attached blood gas analyser.

The study forms an element of the Post Market surveillance plan for the Proxima system and will also generate method comparison data to allow Sphere Medical to submit the Proxima for FDA regulatory clearance.

DETAILED DESCRIPTION:
The PROX006 study is an open and non-randomised study that will be conducted to assess the performance of the Proxima (a CE marked Medical Device)on a wide range of patients with a variety of conditions. This study will allow the performance of the Proxima and the institution's conventional blood gas analyser to be compared when used in the Intensive Care Unit and Operating Theatre.

The PROX006 investigation is an observational method comparison study - the results obtained from the Proxima will be compared with those obtained on the institution's conventional blood gas analyser (BGA). The potential for bias by the user will be negated in this study by directly comparing the results from the BGA and Proxima.

The data/results documented in the Case Report Form (CRF) will be verified during monitoring visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years old
* Patients who have (or will have) an arterial line, which was (will be) inserted for clinical need, will be considered for inclusion in this study
* Patients who give informed consent (or their personal/nominated consultee) to participate in the study
* Patients who are likely to have an arterial line for at least 48 hours.

Exclusion Criteria:

* Patients not indicated or contraindicated for an arterial line
* Refusal of consent by a patient or their personal/nominated consultee to participate
* Not for use with patients with uncorrected hyperphosphataemia, hypocalcaemia or hypercalcaemia.
* The patient is considered by the investigator to be unsuitable for the study

Arterial line location/placement is not dictated by this study, however the following criteria should be considered when deciding if arterial catheter placement is suitable, including but not limited to:

* peripheral vascular disease,
* history of placement site neuropathy or chronic pain,
* history of placement extremity coagulopathy or clot formation,
* history of vascular surgery on same extremity as catheter placement (and/or vascular grafts)
* patients with a plan for perioperative anticoagulation. These patients are at increased risk of known complications such as bleeding and arteriospasm and should be excluded in order to mitigate patient study risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Intensive Care Unit, High Dependency Unit or Operating Theatre who require an arterial line to be inserted as standard care
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
- To obtain quantitative data using patient arterial blood to allow the comparison of Proxima readings with those obtained from a standard commercially available blood gas analyser in a clinical setting. | 4 days for each patient
  Blood gas samples will be analysed on the Proxima and institution's Blood Gas Analyser.
  Additional samples for serum phosphate analysis will be draw and analysed every 24 hours for 3 days.
  1 day follow up period after the Proxima system has been disconnected from the patient

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clutton-Brock, MB ChB FRCA FRCP FFICM, Study Director — Queen Elizabeth Hopsital, Birmingham, UK
Locations (1):
- Queen Elizabeth Hospital, City and Borough of Birmingham, Edgbaston, United Kingdom

REFERENCES:
- See also: Visit above web address more information about this study — http://www.spheremedical.com